CLINICAL TRIAL: NCT06212830
Title: Enhancing Pain Relief After Corneal Collagen Cross-Linking: Exploring New Post-Surgical Treatments
Brief Title: Pain Relief After Corneal Collagen Cross-Linking
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Adi Einan-Lifshitz, Professor, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 177-23
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Provide Evidence-based Recommendations for Clinicians to Optimize Pain Control After CXL
MeSH Terms: interventions — Gabapentin; Anti-Inflammatory Agents, Non-Steroidal; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gabapentin (Active Comparator): This group will receive a combination of drugs including:
  Gabapentin, NSAIDS and Paracetamol.
  Interventions: Drug: Gabapentin; Drug: NSAID; Drug: Paracetamol
- Targin (Active Comparator): This group will receive a combination of drugs including:
  Targin, NSAIDS and Paracetamol.
  Interventions: Drug: Targin; Drug: NSAID; Drug: Paracetamol
- Control (Active Comparator): This group will receive a combination of drugs including:
  NSAIDS and Paracetamol.
  Interventions: Drug: NSAID; Drug: Paracetamol

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 200 mg twice a day, starting from the night prior to the procedure and continue 48 hours after
  Arms: Gabapentin
Drug: Targin — Targin 5 mg twice a day after the procedure for 48 hours
  Arms: Targin
Drug: NSAID — Nurofen (NSAID) 200 mg twice a day after the procedure for 48 hours
Drug: Paracetamol — Paracetamol 500 mg every 4 hours during waking hours after the procedure for 48 hours

SUMMARY:
Keratoconus is a progressive corneal ectasia that can lead to significant visual impairment and decreased quality of life. The introduction of corneal cross-linking (CXL) with riboflavin and ultraviolet-A (UVA) light has revolutionized the treatment of keratoconus by increasing corneal rigidity and arresting disease progression. The epithelium-off protocol, which induces heightened post-surgical discomfort, is the prevailing approach. Despite the success of CXL, postoperative pain is a common side effect that can negatively impact patients' quality of life and impede recovery.

Pain management after CXL is essential for optimizing patient outcomes and satisfaction. Systemic painkillers, though not researched enough, may potentially aid in healing and recovery, minimizing complications and discomfort for the patient.

In this study we will provide evidence-based recommendations for clinicians to optimize pain control after CXL in collaboration with pain specialists.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 15 years
* Patients who are undergoing CXL treatment

Exclusion Criteria:

* Renal and/or hepatic failure
* Patients under the age of 15

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pain questionnaires | The questionnaire will be asked 2, 6, 24 48 and 72 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No